CLINICAL TRIAL: NCT05415228
Title: Expanded Access to Gallium-68 PSMA-11 PET in Patients With Biochemical Recurrent Prostate Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Morand Piert, MD (Other)
Responsible Party: Sponsor-Investigator, Morand Piert, MD, Professor of Radiology, University of Michigan
Organization: University of Michigan (Other)
Other Study IDs: HUM00198146
Record Dates: First submitted 2022-06-02; First posted 2022-06-13 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Prostate Adenocarcinoma
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; N,N'-bis(2-hydroxy-5-(ethylene-beta-carboxy)benzyl)ethylenediamine N,N'-diacetic acid

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — 68Ga-PSMA-11 is a radiopharmaceutical for the detection of prostate cancer using PET/CT imaging
  Other Names: HBED-CC; Glu-urea-Lys(Ahx)-HBED-CC; PSMA-HBED-CC

SUMMARY:
This is an expanded access program using 68Ga PSMA-HBED-CC (68Ga-PSMA-11).

The primary goal of this expanded access program is to make 68Ga PSMA-11 PET/CT imaging available to patients.

DETAILED DESCRIPTION:
Imaging and staging of prostate cancer is critical for surgical and treatment planning. Gallium-68 labeled HBED-CC PSMA (more commonly called 68Ga-PSMA-11) has recently been approved by the FDA for clinical use in a formulation utilized at the University of California in Los Angeles UCLA) and San Francisco (UCSF).

The production process for 68Ga-PSMA-11 at the University of Michigan (UM) is different and not FDA approved. This expanded access program was established to allow a continued use of 68Ga-PSMA-11 produced at the University of Michigan for clinical management for prostate cancer at the University of Michigan.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological proven prostate adenocarcinoma
* Elevated PSA after initial therapy: Post radical prostatectomy (RP) - AUA recommendation. PSA greater than 0.2 ng/mL measured more than 6 weeks after RP and confirmatory persistent PSA greater than 0.2 ng/mL
* Elevated PSA after initial therapy: Post radiation therapy or post focal therapy of prostate gland. Nadir + greater than or equal to 2 ng/mL rise in PSA
* Ability to understand a written informed consent document and the willingness to sign it

Exclusion Criteria:

* Current investigational therapy for prostate cancer
* Unable to lie flat, still, or tolerate a PET/CT scan

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

REFERENCES:
- [Result] Abghari-Gerst M, Armstrong WR, Nguyen K, Calais J, Czernin J, Lin D, Jariwala N, Rodnick M, Hope TA, Hearn J, Montgomery JS, Alva A, Reichert ZR, Spratt DE, Johnson TD, Scott PJH, Piert M. A Comprehensive Assessment of 68Ga-PSMA-11 PET in Biochemically Recurrent Prostate Cancer: Results from a Prospective Multicenter Study on 2,005 Patients. J Nucl Med. 2022 Apr;63(4):567-572. doi: 10.2967/jnumed.121.262412. Epub 2021 Jul 29. PMID 34326126